CLINICAL TRIAL: NCT01391195
Title: Effects of Low Level Laser Therapy (808nm) on Muscle Performance of Young Women Submitted to Physical Training
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Wouber Hérickson de Brito Vieira, Federal University of São Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE - 0100.0.135.000-05
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2005-12

CONDITIONS: Healthy
Keywords: low level laser therapy; muscle performance; fatigue index; endurance training; ventilatory threshold; VO2Max; VO2Peak
MeSH Terms: interventions — Lasers; Laser Therapy; Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser therapy and aerobic capacity (Experimental): Effects of low level laser therapy on aerobic capacity of young women submitted to endurance training
  Interventions: Device: Phototherapy by low level laser therapy

INTERVENTIONS:
Device: Phototherapy by low level laser therapy — Phototherapy by low level laser therapy during 9 weeks
  Other Names: Laser; Laser therapy; Low level laser therapy

SUMMARY:
The study hypothesis is an increase in muscle performance and a higher aerobic adaptation of young women submitted to chronic endurance training program associated to low level laser therapy when compared to chronic aerobic training alone.

DETAILED DESCRIPTION:
The study assessed women muscle performance in isokinetic dynamometry, ventilatory parameters such as ventilatory threshold, VO2Peak, VO2Max, Ventilation. Maximal load in cycle ergometer test (Balke's protocol), Borg Scale and Heart rate were assessed too.

ELIGIBILITY:
Inclusion Criteria:

* healthy young women volunteers
* women with a beginner or moderately trained pattern of physical activity
* body Mass Index (BMI) between 18 and 25kg/m2

Exclusion Criteria:

* previous injury to the femoral quadriceps or hamstrings muscles (within 6 months prior to study)
* osseous or articular disorder in the lower limbs
* cardiovascular system disorders or systemic disease

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2006-01; Primary Completion 2007-04 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Fatigue Index of knee extensor muscles | nine weeks
  Fatigue Index of knee extensor muscles assessed in isokinetic dynamometry.
Ventilatory threshold | nine weeks
  Ventilatory threshold quantified by a gas analyzer.
VO2max | nine weeks
  VO2max quantified by a gas analyzer.
VO2peak | nine weeks
  VO2peak quantified by a gas analyzer.
Maximum load of effort on cycle ergometer (Balke's protocol). | nine weeks
  Maximum load of effort on cycle ergometer quantified in Watts.

SECONDARY OUTCOMES:
Total work of knee extensor muscles | nine weeks
  Total work of knee extensor muscles assessed in isokinetic dynamometry
Peak torque of knee extensor muscles | nine weeks
  Peak torque of knee extensor muscles assessed in isokinetic dynamometry
Borg scale | nine weeks
  Subjective effort perception assessed by Borg scale
Heart rate | nine weeks
  Heart Rate assessed by cardiac frequency meter

CONTACTS AND LOCATIONS:
Overall Officials: Wouber Hérickson B Vieira, PhD, Principal Investigator — Universidade Federal de Sao Carlos; Nivaldo A Parizotto, PhD, Study Director — Universidade Federal de Sao Carlos; Cleber Ferraresi, Ms, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de Sao Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Ferraresi C, de Brito Oliveira T, de Oliveira Zafalon L, de Menezes Reiff RB, Baldissera V, de Andrade Perez SE, Matheucci Junior E, Parizotto NA. Effects of low level laser therapy (808 nm) on physical strength training in humans. Lasers Med Sci. 2011 May;26(3):349-58. doi: 10.1007/s10103-010-0855-0. Epub 2010 Nov 18. PMID 21086010
- [Background] Leal Junior EC, Lopes-Martins RA, de Almeida P, Ramos L, Iversen VV, Bjordal JM. Effect of low-level laser therapy (GaAs 904 nm) in skeletal muscle fatigue and biochemical markers of muscle damage in rats. Eur J Appl Physiol. 2010 Apr;108(6):1083-8. doi: 10.1007/s00421-009-1321-1. Epub 2009 Dec 19. PMID 20024577
- [Background] Lopes-Martins RA, Marcos RL, Leonardo PS, Prianti AC Jr, Muscara MN, Aimbire F, Frigo L, Iversen VV, Bjordal JM. Effect of low-level laser (Ga-Al-As 655 nm) on skeletal muscle fatigue induced by electrical stimulation in rats. J Appl Physiol (1985). 2006 Jul;101(1):283-8. doi: 10.1152/japplphysiol.01318.2005. Epub 2006 Apr 20. PMID 16627677
- [Background] Baroni BM, Leal Junior EC, De Marchi T, Lopes AL, Salvador M, Vaz MA. Low level laser therapy before eccentric exercise reduces muscle damage markers in humans. Eur J Appl Physiol. 2010 Nov;110(4):789-96. doi: 10.1007/s00421-010-1562-z. Epub 2010 Jul 3. PMID 20602109
- [Background] Baroni BM, Leal Junior EC, Geremia JM, Diefenthaeler F, Vaz MA. Effect of light-emitting diodes therapy (LEDT) on knee extensor muscle fatigue. Photomed Laser Surg. 2010 Oct;28(5):653-8. doi: 10.1089/pho.2009.2688. Epub 2010 Jul 13. PMID 20626264
- [Background] Leal Junior EC, Lopes-Martins RA, Baroni BM, De Marchi T, Taufer D, Manfro DS, Rech M, Danna V, Grosselli D, Generosi RA, Marcos RL, Ramos L, Bjordal JM. Effect of 830 nm low-level laser therapy applied before high-intensity exercises on skeletal muscle recovery in athletes. Lasers Med Sci. 2009 Nov;24(6):857-63. doi: 10.1007/s10103-008-0633-4. Epub 2008 Dec 5. PMID 19057981
- [Background] Leal Junior EC, Lopes-Martins RA, Vanin AA, Baroni BM, Grosselli D, De Marchi T, Iversen VV, Bjordal JM. Effect of 830 nm low-level laser therapy in exercise-induced skeletal muscle fatigue in humans. Lasers Med Sci. 2009 May;24(3):425-31. doi: 10.1007/s10103-008-0592-9. Epub 2008 Jul 23. PMID 18649044
- [Background] Leal Junior EC, Lopes-Martins RA, Dalan F, Ferrari M, Sbabo FM, Generosi RA, Baroni BM, Penna SC, Iversen VV, Bjordal JM. Effect of 655-nm low-level laser therapy on exercise-induced skeletal muscle fatigue in humans. Photomed Laser Surg. 2008 Oct;26(5):419-24. doi: 10.1089/pho.2007.2160. PMID 18817474